CLINICAL TRIAL: NCT06352112
Title: Short-term Effects of the Home-Based Hypopressive Exercises in Women With Pelvic Organ Prolapse: A Retrospective Comparative Study
Brief Title: Effects of the Hypopressive Exercises in Women With Pelvic Organ Prolapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: Istanbul Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Turkan Akbayrak, Prof. Dr., Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02.04.2024 - POP
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Pelvic Floor Disorders; Prolapse; Female
MeSH Terms: conditions — Pelvic Floor Disorders; Prolapse

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pelvic Floor Muscle Training (Experimental): Participants received pelvic floor muscle training only.
  Interventions: Other: Pelvic Floor Muscle Training
- Pelvic Floor Muscle Training combined with Hypopressive Exercises (Experimental): Participants received hypopressive exercise in addition to pelvic floor muscle training.
  Interventions: Other: Pelvic Floor Muscle Training; Other: Hypopressive Exercises

INTERVENTIONS:
Other: Pelvic Floor Muscle Training — PFMT consisted of both slow voluntary contractions lasting 15 seconds each (5-s contraction, 5-s hold and 5-s relaxation) and fast voluntary contractions lasting 2-s each. A set of exercises included 10 slow and 10 fast voluntary contractions. During the first week, women performed five sets of exercises a day, and the exercises were continued for eight weeks by increasing five sets each week. The exercises were performed as home exercises.
Other: Hypopressive Exercises — HE program in which different placements of the upper and lower extremities were used in standing, sitting and supine positions, and the participants were asked to perform the exercises with a "hypopressive maneuver" to maintain apnea and rib cage expansion for approximately 10 seconds. Exercises were started with three repetitions a day, and then the number of repetitions was increased to five and/or 10, depending on the participant's tolerance. The exercises were performed as home exercises.
  Arms: Pelvic Floor Muscle Training combined with Hypopressive Exercises

SUMMARY:
The aim of this study was compare home-based pelvic floor muscle training (PFMT) alone and home-based PFMT combined with hypopressive exercise (HE) in terms of pelvic floor muscle (PFM) activation and severity of pelvic floor dysfunction (PFD) in women with pelvic organ prolapse (POP) for eight weeks. For this purpose, the participants were randomly divided into two groups: [PFMT alone (n:15) and PFMT combined with HE(n:17)]. DuoBravo EMG device for evaluation of PFM activation and "Pelvic Floor Distress Inventory-20" was used to evaluate the severity of PFD. All evaluations were performed twice in total, at baseline and at week 8.

DETAILED DESCRIPTION:
Pelvic floor muscle training (PFMT), which provides increased structural support of the pelvic organs by improving the functional strength, endurance and coordination of the pelvic floor muscles (PFM), has been a grade A recommendation based on Level 1 evidence to improve symptoms and stages of pelvic organ prolapse (POP). On the other hand, hypopressive exercises (HE) are a group of exercises that, when applied, relax the diaphragm, activate the abdominal muscles, activate the transversus abdominis muscle by reducing intra-abdominal pressure, thus providing reflex activation in the PFM, and are known to improve urinary incontinence and POP with these features. Although there are studies investigating the effects of both exercise groups on POP, the results of the studies are contradictory and more research is needed on this subject.For this reason, in this study, the investigators aimed to compare home-based PFMT alone and home-based PFMT combined with HE in terms of PFM activation and severity of pelvic floor dysfunction in women with POP for eight weeks.

ELIGIBILITY:
Inclusion Criteria:

* having been diagnosed with POP according to Pelvic Organ Prolapse Quantification System by a gynecologist;
* being literate
* being between 20-50 years

Exclusion Criteria:

* pregnancy;
* having a cooperation problems;
* history of active cancer;
* finding an urinary infection during evaluation;
* being in the menstrual period during the evaluation;
* neurological, orthopedic or serious medical conditions that may affect the patient's pelvic floor functions.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only women with POP were included in the study.
Enrollment: 32 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Pelvic Floor Muscle Activation | at baseline and at week 8
  It was performed with the DuoBravo EMG device. Patients were asked to squeeze the PFM strongly for 5-s and at the end of the contraction, to relax completely by not pushing the perineum downwards for 5-s. This cycle was repeated five times in total, and the muscle activation responses at the end of the measurement were recorded in µV.

SECONDARY OUTCOMES:
Severity of pelvic floor dysfunction | at baseline and at week 8
  It was performed with the "Pelvic Floor Distress inventory-20 (PFDI-20). The total score of the scale is between 0-300 and the higher the score obtained as a result of the survey, the greater the severity of pelvic floor dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Türkan Akbayrak, Prof. Dr., Principal Investigator — Hacettepe University
Locations (1):
- Istanbul Research and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Resende AP, Stupp L, Bernardes BT, Oliveira E, Castro RA, Girao MJ, Sartori MG. Can hypopressive exercises provide additional benefits to pelvic floor muscle training in women with pelvic organ prolapse? Neurourol Urodyn. 2012 Jan;31(1):121-5. doi: 10.1002/nau.21149. Epub 2011 Oct 28. PMID 22038880
- [Result] Bernardes BT, Resende AP, Stupp L, Oliveira E, Castro RA, Bella ZI, Girao MJ, Sartori MG. Efficacy of pelvic floor muscle training and hypopressive exercises for treating pelvic organ prolapse in women: randomized controlled trial. Sao Paulo Med J. 2012;130(1):5-9. doi: 10.1590/s1516-31802012000100002. PMID 22344353
- [Result] Resende APM, Bernardes BT, Stupp L, Oliveira E, Castro RA, Girao MJBC, Sartori MGF. Pelvic floor muscle training is better than hypopressive exercises in pelvic organ prolapse treatment: An assessor-blinded randomized controlled trial. Neurourol Urodyn. 2019 Jan;38(1):171-179. doi: 10.1002/nau.23819. Epub 2018 Oct 12. PMID 30311680
- [Result] Bo K, Angles-Acedo S, Batra A, Braekken IH, Chan YL, Jorge CH, Kruger J, Yadav M, Dumoulin C. Are hypopressive and other exercise programs effective for the treatment of pelvic organ prolapse? Int Urogynecol J. 2023 Jan;34(1):43-52. doi: 10.1007/s00192-022-05407-y. Epub 2022 Nov 23. PMID 36418569
- [Result] Molina-Torres G, Moreno-Munoz M, Rebullido TR, Castellote-Caballero Y, Bergamin M, Gobbo S, Hita-Contreras F, Cruz-Diaz D. The effects of an 8-week hypopressive exercise training program on urinary incontinence and pelvic floor muscle activation: A randomized controlled trial. Neurourol Urodyn. 2023 Feb;42(2):500-509. doi: 10.1002/nau.25110. Epub 2022 Dec 8. PMID 36482844